CLINICAL TRIAL: NCT02500472
Title: Investigation of Kava Effects on the Metabolism of the Tobacco-specific Carcinogen 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK) in Humans
Brief Title: Investigation of Kava Effects on NNK Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015NTLS038
Record Dates: First submitted 2015-06-26; First posted 2015-07-16 (Estimated); Last update posted 2018-04-04 (Actual); Status verified 2017-12

CONDITIONS: Tobacco Smoking
Keywords: Tobacco; Smoking
MeSH Terms: conditions — Tobacco Smoking; Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Kava Supplement (Experimental): See intervention description.
  Interventions: Dietary Supplement: Kava

INTERVENTIONS:
Dietary Supplement: Kava — 3 doses equaling 250 mg kavalactones per day. Participants will take 1 capsule three times daily at 8:00 (± 2 hours), 14:00 (± 2 hours) and 20:00 (± 2 hours) for 7 consecutive days.

SUMMARY:
This is a non-therapeutic, single-arm pilot clinical trial in adult healthy smokers to assess whether kava can alter NNK metabolism in humans.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years
* Current smoker of ≥ 5 cigarettes daily, determined by self-report
* Adequate liver and kidney function, defined as:

  * Bilirubin, alkaline phosphatase, ALT, and AST within normal limits
  * Creatinine <1.2
* Adequate hemoglobin, defined as a hemoglobin ≥12 mg/dL for men and ≥11 for women.
* Ability and willingness to abstain from all medication and dietary supplements for 3 days prior to kava administration, continuing until a minimum of 7 days after kava administration. Topical medications and inhaled medications that do not contain steroids are permitted.
* Ability and willingness to completely abstain from alcohol consumption for 3 days prior to kava administration, continuing until a minimum of 7 days after kava administration
* Ability to understand the investigational nature of the study and provide informed consent
* Willingness to take kava supplement as instructed

Exclusion Criteria:

* Known hepatobiliary disease or impairment
* History of gastric bypass surgery, gastric banding, bowel resection, malabsorption syndromes such as celiac sprue or pancreatic insufficiency, or other conditions that may affect the absorption of kava
* Chronic medication use that cannot be safely stopped
* Use of tobacco products other than cigarettes (i.e. snuff, snuz, smokeless tobacco, cigars, pipes)
* Major or chronic medical medical disease, including heart disease, poorly controlled diabetes, etc., to be adjudicated by the principal investigator
* Women who are pregnant, intend to become pregnant within 3 months of the study period, or who are breastfeeding
* Current or recent (within 12 months) problems with drug use or alcohol dependence by self-report
* Antibiotic use within 2 months of study enrollment by self-report
* Alcohol dependence, abuse, or history of dependence/abuse by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-12-03 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Urinary level (nmol/mL) of total NNAL before and after short-term kava administration | Day 1
  Compare urinary level of total NNAL before and after short-term kava administration
Urinary level (nmol/mL) of total NNAL before and after short-term kava administration | Day 2
  Compare urinary level of total NNAL before and after short-term kava administration
Urinary level (nmol/mL) of total NNAL before and after short-term kava administration | Day 4
  Compare urinary level of total NNAL before and after short-term kava administration
Urinary level (nmol/mL) of total NNAL before and after short-term kava administration | Day 5
  Compare urinary level of total NNAL before and after short-term kava administration
Urinary level (nmol/mL) of total NNAL before and after short-term kava administration | Day 6
  Compare urinary level of total NNAL before and after short-term kava administration
Urinary level (nmol/mL) of total NNAL before and after short-term kava administration | Day 7
  Compare urinary level of total NNAL before and after short-term kava administration

SECONDARY OUTCOMES:
Ratio of urinary NNAL-gluc (nmol/mL) and free NNAL (nmol/mL) before and after short-term kava administration | Day 1
  Compare the ratio of urinary NNAL-gluc and free NNAL before and after short-term kava administration
Ratio of urinary NNAL-gluc (nmol/mL) and free NNAL (nmol/mL) before and after short-term kava administration | Day 2
  Compare the ratio of urinary NNAL-gluc and free NNAL before and after short-term kava administration
Ratio of urinary NNAL-gluc (nmol/mL) and free NNAL (nmol/mL) before and after short-term kava administration | Day 4
  Compare the ratio of urinary NNAL-gluc and free NNAL before and after short-term kava administration
Ratio of urinary NNAL-gluc (nmol/mL) and free NNAL (nmol/mL) before and after short-term kava administration | Day 5
  Compare the ratio of urinary NNAL-gluc and free NNAL before and after short-term kava administration
Ratio of urinary NNAL-gluc (nmol/mL) and free NNAL (nmol/mL) before and after short-term kava administration | Day 6
  Compare the ratio of urinary NNAL-gluc and free NNAL before and after short-term kava administration
Ratio of urinary NNAL-gluc (nmol/mL) and free NNAL (nmol/mL) before and after short-term kava administration | Day 7
  Compare the ratio of urinary NNAL-gluc and free NNAL before and after short-term kava administration
Percentage of subjects experiencing any particular adverse event | Day 4
  Determine the safety of short-term kava administration in healthy smokers
Percentage of subjects experiencing any particular adverse event | Day 7
  Determine the safety of short-term kava administration in healthy smokers
O6-mG adducts level (fmol) in peripheral blood cells before and after short-term kava administration | Day 4
  Quantify O6-mG adducts in peripheral blood cells before and after short-term kava administration
O6-mG adducts level (fmol) in peripheral blood cells before and after short-term kava administration | Day 7
  Quantify O6-mG adducts in peripheral blood cells before and after short-term kava administration

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Fujioka, MD, Principal Investigator — University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Wang Y, Fujioka N, Xing C. Quantitative profiling of cortisol metabolites in human urine by high-resolution accurate-mass MS. Bioanalysis. 2018 Dec;10(24):2015-2026. doi: 10.4155/bio-2018-0182. Epub 2018 Nov 6. PMID 30412681